CLINICAL TRIAL: NCT05295225
Title: Investigating the Analgesic Effects of Green Light Exposure in Normal Human Volunteers
Brief Title: Green Light Exposure in Healthy Volunteers Exposure in Normal Human Volunteers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Mohab Ibrahim, PhD MD, Associate Professor, Anesthesiology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00000370
Record Dates: First submitted 2022-02-22; First posted 2022-03-25 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Light Exposure (Active Comparator): Subjects will complete thermal and mechanical pain threshold detection tests and Electroencephalography (EEG). After completion, subjects will be exposed to a green light-emitting diode for two hours. After exposure, thermal and mechanical pain threshold assessments and Electroencephalography (EEG) will be conducted.
  Interventions: Device: Green Light Emitting Diode
- White Light Exposure (Placebo Comparator): Subjects will complete thermal and mechanical pain threshold detection tests and Electroencephalography (EEG). After completion, subjects will be exposed to a white light-emitting diode for two hours. After exposure, thermal and mechanical pain threshold assessments and Electroencephalography (EEG) will be conducted.
  Interventions: Device: White Light Emitting Diode

INTERVENTIONS:
Device: Green Light Emitting Diode — GLED exposure for two hours
  Other Names: GLED
  Arms: Green Light Exposure
Device: White Light Emitting Diode — WLED exposure for two hours
  Other Names: WLED
  Arms: White Light Exposure

SUMMARY:
This research project is intended to understand the mechanisms of action for the pain-relieving properties of visual green light exposure.

The investigators have shown previously that greenlight exposure decreased acute and chronic pain in both animals and humans. However, the investigators do not yet understand how green light exposure is capable of such function.

DETAILED DESCRIPTION:
Pain is a biological function. There are several pain centers in the brain that modulate the intensity of the pain signal perceived by the brain. Part of the modulations takes place through two separate pathways. The first pathway mediates pain signals and is known as the ascending facilitator pain pathway. The main function of this pathway is to relay the pain signal to the brain to be processed.

The second pathway is known as the descending inhibitory pain pathway. The main function of this pathway is to inhibit the pain signal mediated by the first pathway.

Normal humans typically have a balance between the activities of the ascending and descending pain pathways.

The investigator animal studies suggest that green light therapy exhibits its pain-relieving effects through altering the balance between the ascending and descending pain pathway in a manner to result in an overall reduction or normalization in pain perception.

To test this hypothesis, the investigators propose recruiting 30 healthy human volunteers. The participants will be equally randomized into either green light (treatment) or white light (control) exposure groups. The investigators will initially test the activities of the ascending and descending pathways using thermal and mechanical stimulations. The investigators will also test brain wave activities using a non-invasive EEG device. After establishing the baseline activities of the pain pathways and brain waves, the volunteers will be exposed to the green light or white light at low intensity (4-100 lux) for two hours in our laboratory. After two hours of light exposure, the investigators will again test the activities of the pain pathways using thermal and mechanical stimulation and measure the brain wave EEG activities.

ELIGIBILITY:
Inclusion Criteria:

1. 18-50 years healthy men or women
2. Able to speak and understand English
3. No history of Chronic pain
4. No known neuropathies in areas that testing will take place, (forearms, muscle at the base of thumb on the palm of the hand and upper back/shoulder area.

Exclusion Criteria:

1. Serious mental illness defined as distortions of perception, delusions, hallucinations, and unusual behaviors resulting in loss of contact with reality. This will be assessed during the screening interview.
2. Colorblindness or uncorrected cataracts.
3. Tissue damage in areas that testing will take place, (forearms, muscle at the base of the thumb on the palm of the hand, and upper back/should area.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ascending Pain Pathway | Two hours
  Changes in activity of the ascending pain pathway
Descending Pain Pathway | Two hours
  Changes in activity of the descending pain pathway

SECONDARY OUTCOMES:
Delta Brain Activities | Two hours
  Changes in the baseline of Delta waves of EEG
Theta Brain Activities | Two hours
  Changes in the baseline of Theta waves of EEG
Alpha Brain Activities | Two hours
  Changes in the baseline of Alpha waves of EEG
Sigma Brain Activities | Two hours
  Changes in the baseline of Sigma waves of EEG
Beta Brain Activities | Two hours
  Changes in the baseline of Beta waves of EEG

CONTACTS AND LOCATIONS:
Overall Officials: Mohab Ibrahim, PhD, MD., Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ibrahim MM, Patwardhan A, Gilbraith KB, Moutal A, Yang X, Chew LA, Largent-Milnes T, Malan TP, Vanderah TW, Porreca F, Khanna R. Long-lasting antinociceptive effects of green light in acute and chronic pain in rats. Pain. 2017 Feb;158(2):347-360. doi: 10.1097/j.pain.0000000000000767. PMID 28092651